CLINICAL TRIAL: NCT00557583
Title: A Randomized, Double-blinded, Placebo-controlled, Sequential, Single Ascending Dose Evaluation of the Safety and Pharmacokinetics of VBY-376 in Healthy Adults
Brief Title: Evaluation of Safety and Pharmacokinetics of Single Doses of VBY-376 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virobay Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: VBY-376-001
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Hepatitis C Infection
Keywords: VBY-376 Hepatitis C pharmacokinetics safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: VBY 376 — Doses of 50mg and higher or placebo will be evaluated.

SUMMARY:
The study will evaluate the safety and pharmacokinetics of single doses of VBY-376 in healthy subjects.

DETAILED DESCRIPTION:
Single dose escalation study of 5 dose levels of VBY-376. Eight subjects per group will receive one dose of VBY-376 then have multiple blood draws for pharmacokinetic evaluation and followed for safety with laboratory evaluations, ECG's, vital signs, and adverse events. Safety data will be reviewed before proceeding to the next dose.

ELIGIBILITY:
Inclusion Criteria:

* males and females between 18 and 45 years of age
* screening body mass index between 20 and 29 kg/m2
* in good health with no clinically significant medical conditions
* able to comprehend and willing to sign an informed consent

Exclusion Criteria:

* history of renal, hepatic impairment, stomach or intestinal surgery or resection, malabsorption syndrome
* anemia or blood donation within 8 weeks of check-in
* plasma donation within 4 weeks of check-in
* history of alcoholism or drug addiction within 1 year prior to check-in
* use of drugs of abuse
* no tobacco-containing products within 6 months of study
* participation of any clinical trial within 30 days
* history or presence of abnormal ECG
* no prescription or over-the-counter medications within 14 days of study and during the study
* history of Gilbert's syndrome

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of VBY-376 in single oral doses in healthy subjects. | 7 days

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of VBY-376 after single oral doses and the effect of food on VBY-376. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Flach, MD, Principal Investigator — Covance CRU
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- See also: Sponsor website — http://www.virobayinc.com